CLINICAL TRIAL: NCT04007458
Title: Maine Lung Cancer Coalition: Using CHWs for the Annual Lung Cancer Screening Reminder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Conners (Other)
Responsible Party: Sponsor-Investigator, Anne Conners, Principal Investigator, MaineHealth
Organization: MaineHealth (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1419555
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer
Keywords: Screening
MeSH Terms: conditions — Lung Neoplasms | interventions — College Fraternities and Sororities

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to one of the following two groups:
  1. Control Group:
  o Annual reminder letter only
  1. Intervention Group:
  2. Annual reminder letter and Community Health Worker proactive outreach
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blind to which intervention the subjects have received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Letter (Active Comparator): Patients will receive a letter reminding them that they are overdue for repeat annual screening.
  Interventions: Behavioral: Letter
- Community Health Worker phone call (Experimental): Patients will receive a phone call from community health worker, offering to help them overcome barriers to repeat annual screening and offering to help them schedule their screening.
  Interventions: Behavioral: Community Health Worker Phone Call

INTERVENTIONS:
Behavioral: Letter — MaineGeneral Radiology will generate a reminder letter about their need for an annual low dose CT scan to the subjects in this arm.
  Arms: Letter
Behavioral: Community Health Worker Phone Call — Patients will receive a phone call from community health worker, offering to help them overcome barriers to repeat annual screening and offering to help them schedule their screening.
  Arms: Community Health Worker phone call

SUMMARY:
This research study will test whether support from a Community Health Worker (CHW) to address barriers to annual LDCT screening will result in an increased number of patients who receive the annual screening as per the recommended standard of care compared to passive outreach using a reminder letter.

DETAILED DESCRIPTION:
This research study is a randomized controlled trial comparing phone outreach by a trained Community Health Worker (CHW) following a reminder letter to the reminder letter alone for patients who are at least a month overdue to have a routine annual low dose CT scan (LDCT) screening for lung cancer. CHWs will be able to identify and address barriers to accessing screening for those patients randomized to that arm of the study. Outcomes that will be measured include scheduling and completing the LDCT as well as agreeing to a referral for tobacco treatment.

ELIGIBILITY:
Inclusion Criteria:

* 30 or more pack years of tobacco use
* If no longer using tobacco, no more than 15 years since last use
* At least 13 months since last low dose CT scan screening

Exclusion Criteria:

* Development of serious medical condition that would preclude treatment of lung cancer if found
* Death since baseline screen

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Completed low dose CT scan | through study completion, an average of 1 year
  Percentage of patients who receive low dose CT scan within 3 months of the date on which they were initially contacted by letter

SECONDARY OUTCOMES:
Scheduled low dose CT scan | through study completion, an average of one year
  Percentage of patients who schedule a low dose CT scan within 3 months of the date on which they were initially contacted by letter
Tobacco counseling | through study completion, an average of one year
  Percentage of current smokers in the CHW phone call arm who receive counseling about tobacco treatment
Maine Tobacco Helpline Referral | trhough study compeltion, an average of one year
  Percentage of current smokers in the CHW phone call arm who accept referral to Maine Tobacco Helpline

CONTACTS AND LOCATIONS:
Locations (1):
- MaineGeneral Medical Center, Augusta, Maine, United States